CLINICAL TRIAL: NCT06743555
Title: Surgery After Verifying Existing Disease in Locally Advanced Operable Lung Cancer (SAVED LUNG Study): A Pilot Study
Brief Title: Surgery After Verifying Existing Disease in Locally Advanced Operable Lung Cancer: A Pilot Study
Acronym: SAVED LUNG
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12255
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer; Immunotherapy; Neoadjuvant Therapy; Thoracic Surgery; Complete Response
Keywords: NSCLC; Neoadjuvant immunotherapy; Complete response; Surveillance; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pathologic Complete Response | interventions — Observation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care surgery (Active Comparator): Participants undergo surgery followed by the same surveillance schedule as Arm A. ctDNA testing is conducted 3 weeks post-surgery and again at 6 months. Surveillance includes low-dose CT scans, physical examinations, and ECOG assessments every 3 months for 12 months, with long-term monitoring at regular intervals up to 5 years.
  Interventions: Procedure: Standard-of-care surgery
- Observation without surgery (Experimental): Participants undergo surveillance without surgery, including a low-dose CT scan of the thorax and upper abdomen, ECOG assessment, and physical examination every 3 months for the first 12 months. Additional ctDNA testing is performed 3 weeks post-randomization and at 6 months. Long-term follow-up includes similar assessments every 6-12 months up to 5 years.
  Interventions: Other: Observation without surgery

INTERVENTIONS:
Other: Observation without surgery — Patients randomized to this arm will forego standard-of-care thoracic surgery and will undergo strict surveillance based on serial radiological follow-up and ctDNA monitoring
  Arms: Observation without surgery
Procedure: Standard-of-care surgery — Patients randomized to this arm will undergo standard-of-care thoracic surgery and undergo post-operative surveillance with serial radiological follow-up and ctDNA monitoring
  Arms: Standard-of-care surgery

SUMMARY:
The SAVED LUNG study is a pilot Phase I trial evaluating safety and feasibility of observation versus standard-of-care surgery in operable Stage II-III (excluding N3) NSCLC patients (PD-L1 ≥50%) who achieve complete clinical response following neoadjuvant platinum-doublet chemotherapy and immunotherapy. Participants are randomized to observation or surgery after rigorous restaging, with primary endpoints focusing on safety and feasibility. Secondary objectives include rates of cross-over to surgery, event-free survival, and overall survival, while exploratory endpoints examine ctDNA clearance and its association with clinical response.

DETAILED DESCRIPTION:
After neoadjuvant therapy, all participants undergo intensified re-staging invasive and non-invasive modalities to assess for complete clinical response:

* Chest CT;
* PET/CT scan;
* Bronchoscopy;
* EBUS;
* EUS;
* Re-biopsy of lesions that were deemed to be positive for cancer; this includes re-biopsies of all positive lymph nodes and transthoracic needle aspiration of tumors.

Participants with complete clinical response defined by absence of disease as measured by all the above modalities will be randomized 1:1 to either observation or surgery.

Only patients with complete clinical response will proceed to the randomization stage of the trial. Block randomization will occur 1:1 with two participants per block. All other patients will remain on study and undergo therapy as per standard-of-care and will have follow-up on study. Both groups will have blood collected for ctDNA at this stage. For participants in the surgery arm, the blood sample will be 3 weeks after surgery, while participants in surveillance only arm will have the blood sample 3 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* The participant has provided documented informed consent for the trial.
* Histologically confirmed (by core biopsy) NSCLC and confirmed clinical stages II-III (excluding N2) NSCLC (AJCC 8th edition) amenable to receive neoadjuvant chemo-immunotherapy defined by: nivolumab 3mg/kg Q3W in combination with platinum doublet chemotherapy (cisplatin or carboplatin with paclitaxel or pemetrexed Q3W) for 3 cycles.
* PD-L1 tumor proportion score >50%
* Has no history of immunodeficiency, HBV, HCV, HIV.
* For female participants:

  1. Has no active pregnancy (Refer to "Female participants").
  2. For a woman of child-bearing potential (WOCBP), use of a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) during the intervention period and for at least 180 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period.
  3. A WOCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within either 24 hours (urine) or 72 hours (serum) before the first dose of study intervention.
  4. If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has adequate hematological, renal and hepatic function per Investigator discretion required for platinum-doublet chemotherapy plus immunotherapy.
* Has signed the written consent.

Exclusion Criteria:

* Has one of the following tumor locations/types:

  1. NSCLC involving the superior sulcus
  2. Large cell neuro-endocrine cancer (LCNEC)
  3. Sarcomatoid tumor
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has had an allogenic tissue/solid organ transplant.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
* Has a known additional malignancy that is progressing or requires active treatment within the past (5 years). Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, bladder carcinoma, or carcinoma in situ (eg, in situ cervical cancer or breast carcinoma) that have undergone potentially curative therapy are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Safety | From randomization through 5 years of follow-up
  Adverse events will be determined as type and grade using the CTCAE v5.0.
Feasibility | First two years of the study
  Recruitment rate will be defined as the total number of patients recruited (consented) out of the total number of patients approached.

SECONDARY OUTCOMES:
Complete clinical response | Restaging 3 weeks after completion of neoadjuvant therapy (3 cycles of nivolumab and platinum-doublet chemotherapy)
  Defined by absence of cancer in all of the following evaluations:
  * Chest CT;
  * PET/CT scan;
  * Bronchoscopy;
  * EBUS;
  * EUS;
  * Re-biopsy of lesions that were deemed to be positive for cancer; this includes re-biopsies of all positive lymph nodes and transthoracic needle aspiration of tumors.
Cross-over to surgery | From randomization through 5 years of follow-up
  Defined as occurrence of surgery for lung cancer in the observation arm
Event-free survival (EFS) at 12 months | 12 months following randomization
  Defined as the proportion of patients remaining event-free at 12 months, from the time of randomization. Patients who are alive without a documented progression will be censored at the time of their last disease evaluation.
Overall survival (OS) at 12 months | 12 months following randomization
  Defined as the proportion of patients alive at 12 months, from the time of randomization.
Circulation tumor DNA (ctDNA) clearance | 3 weeks post-randomization (surveillance arm) or 3 weeks post-surgery (standard-of-care surgery arm)
  Defined as presurgery change from detectable levels of ctDNA before cycle 1 to undetectable ctDNA before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Desilets, MD, MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848